CLINICAL TRIAL: NCT04154462
Title: Evaluation of the Use of Medical Scribes on Provider Efficiency, Patient Satisfaction, and Wait Times in VAMC Emergency Departments and Specialty Care Clinics
Brief Title: Evaluation of the Use of Medical Scribes in VAMC Emergency Departments and Specialty Care Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Garrido, Associate Director, VA Boston Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PEPReC Protocol #2019-001; VA QUERI PEC #16-001 (Other Grant/Funding Number: VA QUERI)
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Medical Scribes
Keywords: workforce; medical records; documentation; efficiency; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: A two-arm randomized field experiment is being used to assess the effect of medical scribes on productivity, wait times, and patient satisfaction. OVAC will work with participating VAMCs to identify providers to participate in the pilot. A varied provider pool will limit selection bias but must be balanced with recruitment and retention of providers. The goal is to keep the provider-scribe pairs consistent throughout the pilot.
  Each VAMC site randomized to treatment will have two VA employee scribes and two contract scribes. Two medical scribes, ideally one employee and one contract, will be assigned to one physician, with two physicians and/or Licensed Independent Practitioners (LIP) participating at each facility. Scribes will work with others if the provider partner is not available during a scheduled shift. Power analyses have been conducted to determine the minimum effect size for each outcome with 80% power, which will be useful for putting the final results into context.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): The VAMC sites randomized to the comparison arm will not have medical scribes introduced into emergency departments or specialty clinics.
- Treatment (Experimental): The VAMC sites randomized to the treatment arm are each expected to have four medical scribes, with two being VA employees and two being contractors, introduced into emergency departments or specialty clinics to assist providers during patient encounters.
  Interventions: Other: Scribes

INTERVENTIONS:
Other: Scribes — Section 507 of the MISSION Act of 2018 mandates a two-year pilot of medical scribes in VA specialty clinics and emergency departments. Medical scribes assist health care providers by helping to administratively expedite an episode of care through the recording of patient information and updating patient records. Scribes are trained but non-licensed professionals, often deployed in emergency departments and outpatient clinic settings, that observe and document patient encounters but do not participate in clinical care.
  Arms: Treatment

SUMMARY:
Background and study aims: Medical scribes are trained paraprofessionals that assist providers with documenting patient encounters. Prior evidence suggests that scribes may be effective in increasing provider productivity and satisfaction, and decreasing provider time spent on documentation without negatively affecting patient satisfaction. Section 507 of the MISSION Act of 2018 mandated a two-year pilot of medical scribes, which will begin in March 2020 in specialty clinics and emergency departments (EDs) of twelve VA Medical Centers (VAMCs) across the country. The aims of this study are to understand how the introduction of scribes and scribe training affect provider efficiency, patient and provider satisfaction, wait times, and daily patient volume in the VA context.

Who can participate? Urban and rural VAMCs willing to be assigned medical scribes for use in EDs or selected high wait time specialty clinics (cardiology, orthopedics).

What does the study involve? Four medical scribes will be assigned to each of the 12 VAMC sites randomized into treatment with the VA hiring half as new employees and contracting out for the remaining half. 30% of the scribes will be assigned to emergency departments and the other 70% will be assigned to specialty care. Remaining sites that expressed interest in the pilot but were not randomized treatment will be used as comparators. Provider productivity, patient volume, wait times, and patient satisfaction from the treated sites will be compared to baseline (pre-scribe) data as well as data from comparison sites.

What are the possible benefits and risks of participating? VAMCs where medical scribes are introduced may see gains in provider efficiency, reduced wait times, and increased patient satisfaction due to the shifting of administrative burdens associated with documenting patient encounters in electronic health records from providers to these trained professionals. The introduction of medical scribes could complicate patient encounters by making some patients and/or providers uncomfortable.

Where is the study run from? This study is being coordinated by the Partnered Evidence-based Policy Resource Center (PEPReC) at the VA Boston Healthcare System in collaboration with the VA Office of Veterans Access to Care (OVAC).

When is the study starting and how long is it expected to run for? March 2020 to February 2022

Who is funding the study? U.S. Veterans Health Administration

ELIGIBILITY:
Inclusion Criteria:

• Expression of interest by VAMC

Exclusion Criteria:

• Lack of appropriate site capabilities

The VA Office of Veterans Access to Care developed a list of 32 interested VAMCs based on email surveying, which were categorized based on location (urban, rural), desired scribe deployment (ED, specialty care), and underserved (based on high new patient specialty care wait times). 12 VAMCs were then randomly selected for the treatment, accounting for the requirements of the law, OVAC preferences, and site capabilities, with the remainder used as comparison sites.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Pay period work relative value-based provider efficiency | Approximately 42 months
  Pay period work relative value-based provider efficiency is measured using administrative data collected by the VA Corporate Data Warehouse in pay period increments
Pay period visit-based provider efficiency | Approximately 42 months
  Pay period visit-based provider efficiency is measured using administrative data collected by the VA Corporate Data Warehouse in pay period increments
Daily visit-based provider efficiency | Approximately 42 months
  Daily visit-based provider efficiency is measured using monthly-based provider efficiency, scaled by full-time-equivalent days; this is based on administrative data collected by the VA Corporate Data Warehouse in pay period increments
Days to completed consult | Approximately 42 months
  Days to completed consult is measured using administrative data collected by the VA Corporate Data Warehouse in pay period increments
Days to scheduled consult | Approximately 42 months
  Days to scheduled consult is measured using administrative data collected by the VA Corporate Data Warehouse in pay period increments
Unique patient volume | Approximately 42 months
  Unique patient volume is measured using administrative data collected by the VA Corporate Data Warehouse in pay period increments
Patient satisfaction | Approximately 42 months
  Patient satisfaction is measured using V-Signals survey data collected by the VA Office of Veterans Experience in pay period increments

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pizer, PhD, Principal Investigator — Boston VA Healthcare System
Locations (12):
- United States (12):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Togus VA Medical Center, Augusta, Maine
  - Fort Harrison VA Medical Center, Helena, Montana
  - Manchester VA Medical Center, Manchester, New Hampshire
  - East Orange VA Medical Center, East Orange, New Jersey
  - Fargo VA Medical Center, Fargo, North Dakota
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma
  - Audie L. Murphy VA Hospital, San Antonio, Texas
  - Olin E. Teague Veterans' Medical Center, Temple, Texas
  - Hampton VA Medical Center, Hampton, Virginia
  - Louis A. Johnson VA Medical Center, Clarksburg, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearson, E., Frakt, A., & Pizer, S. (2018, December). Medical Scribes, Productivity, and Satisfaction. Partnered Evidence-based Policy Resource Center Policy Brief, 3(2).
- [Derived] Palani S, Saeed I, Legler A, Sadej I, MacDonald C, Kirsh SR, Pizer SD, Shafer PR. Effect of a National VHA Medical Scribe Pilot on Provider Productivity, Wait Times, and Patient Satisfaction in Cardiology and Orthopedics. J Gen Intern Med. 2023 Jul;38(Suppl 3):878-886. doi: 10.1007/s11606-023-08114-6. Epub 2023 Jun 20. PMID 37340268
- See also: S.2372 - VA MISSION Act of 2018 — https://www.congress.gov/bill/115th-congress/senate-bill/2372/text